CLINICAL TRIAL: NCT04200846
Title: Frailty in Liver Transplant Exercise (FLEX) Trial
Acronym: FLEX
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Jonathan Stine, Assistant Professor of Medicine & Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00014084
Record Dates: First submitted 2019-12-11; First posted 2019-12-16 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Frailty; Liver Transplants
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: An interventional pilot trial will be performed with 21 randomized subjects who are aged 18-75 years who are frail according to the LFI to a 3-month exercise intervention (n=14) versus standard of care (n=7) with no change in activity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise intervention (Experimental): Private supervised strength training exercise (e.g., body weight or dumbbell exercises) will occur in the Cancer Center Exercise Medicine Unit or the Hershey Center for Applied Research (HCAR) two days a week. In addition, subjects will be instructed to exercise on their own, at home, three days a week doing 30 minutes of moderate intensity aerobic exercise (e.g., walking at 45-55% maximum heart rate determined by the formula max heart rate = 220bpm - 0.64*age in years).
  Interventions: Behavioral: Exercise intervention
- Control (No Intervention): Subjects in the control condition will be instructed to continue their medical care at the discretion of their treating medical professional and to maintain their current exercise level. Weekly phone calls will be performed to ensure adherence to the protocol (no changes in activity). Subjects will report to Penn State on a monthly basis for interim history and physical to confirm self-reports. Subjects will also be given a FitBit ChargeHR3 and downloaded data review will be performed monthly at the in-person visits.

INTERVENTIONS:
Behavioral: Exercise intervention — Subjects in this group will be asked to exercise 5 days a week. Two days on-site with an Exercise Physiologist and the other 3 days at home.
  Arms: Exercise intervention

SUMMARY:
Frailty is common in patients with end-stage liver disease. It's characterized by reduced strength, low endurance and reduced physical function. While exercise intervention can improve frailty in geriatric patients without liver disease, whether or not exercise intervention can improve frailty in liver transplant candidates remains unknown.

DETAILED DESCRIPTION:
The long-term goal is to better understand how exercise impacts frailty in order to identify treatments that can improve both patient-oriented outcomes and access to liver transplantation for end-stage liver disease patients. The specific objective of this proposal is to generate pilot feasibility data required for future multicenter R01 application to the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) which will test the novel central hypothesis that exercise improves frailty and lessens waiting-list mortality. Additionally, another goal of the study is to establish an optimal frailty tool for liver transplant candidates.

ELIGIBILITY:
Inclusion Criteria:

* Adults age ≥18 or ≤75 years
* Frail as defined by a LFI score of >4.5
* Under evaluation or listed for liver transplant

Exclusion Criteria:

* Active cardiac symptoms (e.g., chest pain, shortness of breath at rest, palpitations)
* Positive response to Get Active Questionnaire (GAQ) (validated activity questionnaire that indicates if exercise is unsafe)
* Institutionalized/prisoner
* Severe medical comorbidities/psychiatric illness at the discretion of the Study Principal Investigator (PI)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants able to complete the trial | up to 52 weeks
  Defined as 50% of subjects completing >80% of the sessions.
Incidence of Treatment-Emergent Adverse Events as assessed by GCP guidelines | up to 52 weeks
  This study aims to examine the incidence of adverse events. If exercise in frail liver transplant candidates is safe. 5% serious adverse events or fewer will deem the trial as safe. If more than 5% serious adverse events occur, the trial is determined to be unsafe.
Rate of enrollment | up to 52 weeks
  Net enrollment rates, which are calculated by dividing the number of subjects approached by the number of subjects that enroll in the trial. The work with the ongoing NASHFit and completed ENACT Trials and the work of others performing exercise-based trials in patients with cirrhosis(50) has established >50% enrollment of subjects approached as a threshold of acceptability.

IPD SHARING:
Plan to Share IPD: No